CLINICAL TRIAL: NCT03388138
Title: Clinical Evaluation of Etafilcon A With Ketotifen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR-5930
Record Dates: First submitted 2017-12-22; First posted 2018-01-02 (Actual); Results first posted 2021-03-16 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Visual Acuity
MeSH Terms: interventions — Ketotifen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- K-Lens (Active Comparator): etafilcon A with ketotifen. Subjects between the ages of 18-40 will be randomized into the K-Lens arm and will be scheduled for a total of two study visits with approximately 6-9 days in between.
  Interventions: Combination Product: etafilcon A with ketotifen
- Placebo Contact Lens (Placebo Comparator): 1-Day Acuvue. Subjects between the ages of 18-40 will be randomized into the Placebo arm and will be scheduled for a total of two study visits with approximately 6-9 days in between.
  Interventions: Device: 1-Day ACUVUE

INTERVENTIONS:
Combination Product: etafilcon A with ketotifen — Etafilcon A with ketotifen
  Arms: K-Lens
Device: 1-Day ACUVUE — 1-Day ACUVUE
  Arms: Placebo Contact Lens

SUMMARY:
This clinical study is a randomized, double-masked, bilateral, controlled, two-arm parallel group, multi-site, 1-Week, 2-visit dispensing study. Subjects between the ages of 18-40 will be randomized into a placebo arm or an investigational K-Lens arm.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Between 18 and 39 (inclusive) years of age at the time of baseline visit.
  4. The subject must be a habitual lens wearer for a least 6 days/week and for a minimum of 8 hours per day over the last month.
  5. The subject's contact lens correction must be in the range of -1.00 D to -6.00 D (inclusive) in each eye.
  6. The subject's refractive cylinder must be 1.00 D or less in each eye.
  7. Have a spherocylindrical best corrected visual acuity of 20/30 or better in each eye (Snellen Visual Acuity).

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating.
  2. Any systemic disease (e.g., Sjögren's Syndrome), allergies, infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g. rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with contact lens wear and/or participation in the study.
  3. Use of systemic medications (e.g., chronic steroid use) that are known to interfere with contact lens wear.
  4. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion.
  5. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear, history of strabismus, or current monovision, multi-focal, or toric contact lens correction.
  6. Any current use of rewetting drops or ocular medication.
  7. Any previous, or planned (during the course of the study) ocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.).
  8. Any grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA Biomicroscopy Scale.
  9. Any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that would contraindicate contact lens wear.
  10. Any known hypersensitivity or allergic reaction to ketotifen.
  11. Participation in any eye drop, contact lens or lens care product clinical trial within 14 days prior to study enrollment.
  12. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 143 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2018-02-09 (Actual); Study Completion 2018-02-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Vue Optical Boutique, Jacksonville, Florida
  - Maitland Vision Center, Maitland, Florida
  - St. Lucy's Vision Center, Tampa, Florida
  - Kannarr Eye Care, Pittsburg, Kansas
  - Sacco Eye Group, Vestal, New York
  - Botetourt Eyecare, LLC, Salem, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 143 subjects were enrolled into this study. Of those enrolled, 141 were dispensed a study lens and 2 subjects were enrolled but not dispensed. Of the dispensed subjects 140 completed the study and 1 discontinued from the study.
Groups:
- Etafilcon A With Ketotifen: Subjects that were randomized to the etafilcon A with ketotifen contact lens throughout the entire duration of the study.
- Etafilcon A: Subjects that were randomized to the etafilcon A contact lens throughout the entire duration of the study.
Period: Overall Study
Arm/Group | Etafilcon A With Ketotifen | Etafilcon A
Started | 94 | 47
Completed | 93 | 47
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: All subjects that were dispensed a study lens.
Groups:
- Total: Total of all reporting groups
Arm/Group | Etafilcon A With Ketotifen | Etafilcon A | Total
Number analyzed (Participants) | 94 | 47 | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (4.98) | 29.6 (4.56) | 30.1 (4.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 31 | 90
  Male | 35 | 16 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 1 | 5
  Black or African American | 7 | 3 | 10
  White | 83 | 43 | 126
Region of Enrollment [Number; unit: participants]
  United States | 94 | 47 | 141

OUTCOME MEASURES:

1. Primary Outcome: Monocular Contact Lens-corrected Distance Visual Acuity (Per-Protocol Population)
Description: Monocular contact lens-corrected distance visual acuity was assessed using a logMAR visual acuity scale. This was evaluated for each eye, under high luminance and high contrast conditions at 4 meters from ETDRS charts. Distance visual acuity was reported by lens type and visit.
Time Frame: Baseline (Visit 1) and 1-week follow up (Visit 2)
Population: Per-protocol (PP) population which consists of all subjects who completed the study without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Groups:
- Etafilcon A With Ketotifen: Subjects that wore the etafilcon A with ketotifen contact lens throughout the entire duration of the study.
- Etafilcon A: Subjects that wore the etafilcon A contact lens throughout the entire duration of the study.
Arm/Group | Etafilcon A With Ketotifen | Etafilcon A
Number analyzed (Participants) | 93 | 46
Number analyzed (eyes) | 186 | 92
logMAR
  Visit 1 (Baseline) | -0.111 (0.0702) | -0.109 (0.0809)
  Visit 2 (1-week follow up) | -0.115 (0.0717) | -0.118 (0.0814)
Statistical Analysis 1: Comparison: Etafilcon A With Ketotifen vs Etafilcon A; Test type: Non-Inferiority — Non-inferiority of the etafilcon A with ketotifen lens relative to the etafilcon A lens was established if the upper limit of the 95% confidence interval was below 0.1 logMAR; Linear Mixed Model; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least-Square Mean Difference = 0.0017, 95% CI 2-sided [-0.021 to 0.025], Standard Error of Mean 0.01169 — LS Mean difference was calculated as etafilcon A with ketotifen - etafilcon A

2. Primary Outcome: Monocular Contact Lens-corrected Distance Visual Acuity (Modified Intent-to-Treat Population)
Description: as for outcome 1
Time Frame: Baseline (Visit 1) and 1-week follow up (Visit 2)
Population: Modified intent-to-treat (MITT) which consists of all the subjects who were administered either study lens excluding subjects who drop out prior to administering any study article.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Etafilcon A With Ketotifen | Etafilcon A
Number analyzed (Participants) | 94 | 47
Number analyzed (eyes) | 188 | 94
logMAR
  Visit 1 (Baseline) | -0.109 (0.0740) | -0.110 (0.0806)
  Visit 2 (1-week follow up) | -0.115 (0.0717) | -0.117 (0.0815)
Statistical Analysis 1: Comparison: Etafilcon A With Ketotifen vs Etafilcon A; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Linear Mixed Model; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least-Square Mean Difference = 0.0007, 95% CI 2-sided [-0.022 to 0.024], Standard Error of Mean 0.01158 — LS Mean difference was calculated as etafilcon A with ketotifen - etafilcon A

3. Secondary Outcome: The Number of Eyes With Clinically Significant Slit Lamp Findings
Description: Slit lamp findings were assessed using a biomicroscope for each subject eye at all scheduled and unscheduled visits. Clinical significant slit lamp findings are defined as Grade 3 or Grade 4. (Grade 0=None, Grade 1=Trace, Grade 2=Mild, Grade 3=Moderate and Grade 4= Severe). The data was dichotomized as 1=Grade 3 or Grade 4 and 0, otherwise. The number of eyes with clinically significant slit lamp findings for each lens type was reported.
Time Frame: Up to 1-Week Follow-up
Population: Modified intent-to-treat (MITT) which consists of all the subjects who were administered either study lens excluding subjects who drop out prior to administering any study article. MITT is identical to safety population.
Measure: Number; unit: Number of Eyes
Units Other Than Participants: eyes
Arm/Group | Etafilcon A With Ketotifen | Etafilcon A
Number analyzed (Participants) | 94 | 47
Number analyzed (eyes) | 188 | 94
Number of Eyes | 0 | 0

4. Secondary Outcome: The Number of Eyes With Unacceptable Lens Fitting
Description: Lens fit was assessed for each subject and eye using a biomicroscope. Unacceptable lens fit was assessed at all scheduled and unscheduled visits. A subject was deemed to have an unacceptable lens fitting if they met any of the following criteria: (1) Limbal exposure at primary gaze with extreme eye movement, (2) edge lift, (3) excessive movement in primary up gaze, (4) insufficient movement in all three of the following conditions: primary gaze, up gaze and push up test. The number of eyes with unacceptable lens fitting was reported for each lens type.
Time Frame: Up to 1-Week Follow-up
Population: as for outcome 3
Measure: Number; unit: eyes
Units Other Than Participants: Number of Eyes
Arm/Group | Etafilcon A With Ketotifen | Etafilcon A
Number analyzed (Participants) | 94 | 47
Number analyzed (Number of Eyes) | 188 | 94
eyes | 0 | 1

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Approximately 1-Week per subject.
Description: All subjects dispensed at least 1 study lens.
Arm/Group | Etafilcon A With Ketotifen | Etafilcon A
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/47
Other Adverse Events (participants affected / at risk) | 0/94 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/38/NCT03388138/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-29): https://cdn.clinicaltrials.gov/large-docs/38/NCT03388138/SAP_001.pdf